CLINICAL TRIAL: NCT04110704
Title: An Investigation Into the Role of Previous in Labour Caesarean Section in Future Preterm Birth Risk and Management Strategies
Brief Title: Cerclage After Full Dilatation Caesarean Section
Acronym: CRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 261294; 42833 (Other: CPMS)
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Preterm Birth; Preterm Premature Rupture of Membrane; Preterm Spontaneous Labor With Preterm Delivery
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transvaginal cerclage (Active Comparator)
  Interventions: Procedure: Insertion of transvaginal cerclage
- Active monitoring (No Intervention)

INTERVENTIONS:
Procedure: Insertion of transvaginal cerclage — Transvaginal cerclage is inserted in women with a high risk of preterm birth. However it is unknown whether this alongside cervical length monitoring improves the incidence of preterm birth. The cerclage is inserted under regional analgesia.
  Arms: Transvaginal cerclage

SUMMARY:
CRAFT-OBS: Observational Study; To evaluate subsequent pregnancy risk of preterm birth in women with a history of previous caesarean in established labour. This prospective study using clinically acquired cervical length and quantitative fetal fibronectin data will help establish a predictive model of preterm birth <34 weeks and <37 weeks.

CRAFT-RCT: Randomised controlled trial arm; To assess treatment for short cervix in women at high risk of preterm birth following a caesarean section at full dilatation

CRAFT-IMG: Imaging sub-study; To aid understanding of micro and macrostructural features within the cervix which predisposes to preterm birth in women with a previous full dilatation caesarean section. This will use MRI and an advanced transvaginal ultrasound protocol and to assess if structural changes can be visualised in the cervix.

ELIGIBILITY:
CRAFT-OBS

Inclusion Criteria:

* Pregnant women under 23+6 weeks gestation with a history of previous caesarean section in labour.
* Singleton pregnancy.
* Willing and able to give informed consent (with or without interpreter).

Exclusion Criteria:

* Under 16 years of age.
* Inability to give informed consent.
* Previous caesarean section carried out before labour.
* Women who have been commenced on management with progesterone, a cerclage or arabin pessary as part of their care or another research study

CRAFT-RCT:

Inclusion criteria:

* Pregnant women up to 23+6 weeks gestation with a history of FDCS.
* Short cervix (<=25mm) on transvaginal ultrasound scan.

Exclusion criteria:

* Women with persistent fresh vaginal bleeding evident on speculum examination.
* Women with visible fetal membranes evident on speculum examination or open cervix on ultrasound scan.
* Women with severe abdominal pain/evidence of sepsis (as judged by attending clinician).
* Known significant congenital or structural or chromosomal fetal abnormality.
* Suspected or proven rupture of the fetal membranes at the time of recruitment.

CRAFT-IMG

Inclusion criteria:

* Pregnant women between 14+0 and 23+6 weeks gestation with a history of FDCS.

Exclusion criteria:

* Contraindications to MRI, e.g. claustrophobia, BMI >40 kg/m2 (due to technical limitations of scanner) or a women with a non-MRI compatible metallic implant.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
CRAFT-OBS: Number of participants with spontaneous preterm birth rate < 37 weeks gestation | Up to 42 weeks
CRAFT-RCT: Number of participants with spontaneous preterm birth <34 weeks gestation | Up to 42 weeks

SECONDARY OUTCOMES:
CRAFT-OBS: Short-term pregnancy and neonatal outcomes, including a composite of neonatal death and morbidity. | Up to 48 weeks
  We will assess the number of antepartum/intrapartum stillbirths plus neonatal deaths prior to discharge from neonatal services.
CRAFT-OBS: Number of participants with adverse perinatal outcome, defined as a composite outcome of death (antepartum/intrapartum stillbirths plus neonatal deaths prior to discharge from neonatal services) | Up to 48 weeks
CRAFT-OBS: Number of participants who deliver <34 weeks gestation | Up to 42 weeks
CRAFT-OBS: Gestation at delivery | Up to 42 weeks
  The proportion of participants who delivery at each gestation of completed weeks
CRAFT-OBS: Late miscarriage (14+0-23+6 weeks) rate | Up to 42 weeks
CRAFT-OBS: Any cervical length measurements taken antenatally | Up to 42 weeks
CRAFT-OBS: Number of antenatal hospital appointments | Up to 42 weeks
CRAFT-OBS: Number of hospital admissions | Up to 42 weeks
CRAFT-OBS: cervicovaginal fetal fibronectin protein levels taken at any gestation if taken | Up to 42 weeks
CRAFT-OBS: Number of ultrasound indicated antenatal interventions | Up to 42 weeks
CRAFT-OBS: Predictive modelling (QUIPP app) to evaluate the ability of CL and fFN to determine risk of preterm birth <34 and <37 weeks | Up to 42 weeks
CRAFT-OBS: Number of participants with other maternal and fetal morbidities, as per COPOP core outcome set for preterm birth intervention studies | Up to 48 weeks
  COPOP core outcomes
CRAFT-RCT: Number of participants with an adverse perinatal outcome | Up to 48 weeks
CRAFT-RCT: Gestation at delivery | Up to 42 weeks
  Proportion of participants who deliver at each gestation of completed weeks
CRAFT-RCT: Number of women needing insertion of a rescue cerclage (done when membranes exposed or bulging) | Up to 30 weeks
CRAFT-RCT: Time between intervention and delivery. | Up to 42 weeks
CRAFT-RCT - Health costs at 28 days post-delivery. | Up to 48 weeks
CRAFT-IMG: Evidence of cervical injury | Up to 40 weeks
  Size of any cervical lesion and its location seen on MRI or ultrasound scans

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: IRAS 261294 — http://preview-kcl.cloud.contensis.com/Preview/1/research/project?id=478a6e61-4446-4a12-945e-c41a3879371d

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT04110704/Prot_SAP_000.pdf